CLINICAL TRIAL: NCT02365038
Title: ART-2 Pilot: A Controlled, Randomized Trial to Assess the Feasiblity of a Driving Pressure Limited Ventilation vs. Standard Strategy (ARDSNet) in Patients With ARDS
Brief Title: ART-2 Pilot - Driving Pressure Limited Ventilation for Patients With ARDS
Acronym: ART2pilot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART2pilot
Record Dates: First submitted 2015-02-06; First posted 2015-02-18 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2015-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Driving pressure limited ventilation (Experimental): Driving pressure limited ventilation
  Interventions: Other: Driving pressure limited ventilation
- Conventional ventilation (Active Comparator): Mechanical ventilation as proposed in the ARDSNet protocol.
  Interventions: Other: Conventional ventilation

INTERVENTIONS:
Other: Driving pressure limited ventilation — We will use volume controlled ventilation or pressure support in the weaning phase. We will adjust tidal volume between 3 and 8 mL/Kg of predicted body weight in order to achieve a driving pressure of 13 cmH2O. The respiratory rate will be titrated to achieve a pH between 7.30 and 7.45 (maximum respiratory rate is 50 breathings per minute). We will not limit plateau pressure in this arm.
  Arms: Driving pressure limited ventilation
Other: Conventional ventilation — ARDSNet Strategy: conventional mechanical ventilation strategy with tidal volume between 4 and 6 mL/kg of predicted body weight and plateau pressure limited to 30 cmH2O.
  Other Names: ARDSNet strategy
  Arms: Conventional ventilation

SUMMARY:
This is a multicenter randomized controlled pilot trial to investigate the feasibility of a driving pressure limited mechanical ventilation strategy compared to the ARDS Clinical Network strategy (conventional strategy) in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Mechanical ventilation has the potential to produce or worsen alveolar injury. Driving pressure is the difference between plateau pressure and PEEP. Evidence from observational studies suggests that elevated driving pressure is the main independent determinant of ventilator-induced lung injury, however clinical trials are needed to establish whether targeting low driving pressures can improve clinical outcomes in patients with acute respiratory distress syndrome (ARDS). Thus, ART2pilot is a multicenter randomized controlled trial to assess the feasibility of a driving pressure limited mechanical ventilation strategy compared to the ARDS Clinical Network strategy (conventional strategy) in patients with ARDS. Patients considered to this trial are those in mechanical ventilation with diagnosis of ARDS of less than 72 hours duration. We will exclude patients with less than 18 years old; contraindication to hypercapnia such as intracranial hypertension or recent acute coronary syndrome; patients in which a high probability of death within 24 hours is anticipated and patients under exclusive palliative care. Eligible patients will be randomized to the driving pressure limited ventilation strategy or ARDSNet strategy. The primary outcome is driving pressure between days 1 and 3.

ELIGIBILITY:
Inclusion criteria:

* Patients on invasive mechanical ventilation with diagnosis of ARDS of less than 72 hours duration.

Exclusion criteria:

* Less than 18 years old.
* Presence of any contraindication to hypercapnia as suspected or confirmed intracranial hypertension or recent (<7 days) acute coronary syndrome.
* Patients in which a high probability of death within 24 hours is anticipated.
* Patients under exclusive palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06-12 (Actual); Primary Completion 2017-02-25 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Mean driving pressure between day 1 and day 3 | Day 1 to Day 3 after randomization
  Driving pressure is the difference between plateau pressure and PEEP. It will be measured every morning in patients without spontaneous efforts. As every patients will have up to three measurements, we will consider the mean driving pressure for each patient.

SECONDARY OUTCOMES:
Adherence to study procedures: daily adjustement of driving pressure in experimental group and tidal volume in the control group | Days 1 to 7
Rate of driving pressure equal or lower than 13cmH2O | Days 1 to 3 after randomization
Mean PEEP from day 1 to 7 | Days 1 to 7
Mean tidal volume from day 1 to day 7 | Days 1 to 7
Mean static compliance of the respiratory system from day 1 to day 7 | Days 1 to 7
Mean plateau pressure from day 1 to day 7 | Days 1 to 7
Mean driving pressure from day 1 to day 7 | Days 1 to 7
Mean respiratory rate from day 1 to day 7 | Days 1 to 7
Barotrauma | Days 1 to 7
Severe acidosis (pH <7.1) | Days 1 to 7
Other adverse events | Days 1 to 7
Length of stay in intensive care unit | ICU stay
Length of stay in hospital | In-hospital stay
Mechanical ventilation free days from day 0 to day 28 | From day 0 to day 28
ICU mortality | ICU stay
In-hospital mortality | Hospital stay
28-day survival | From day 0 to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, PhD, Study Chair — Hospital do Coracao (Heart Hospital)

REFERENCES:
- [Derived] Pereira Romano ML, Maia IS, Laranjeira LN, Damiani LP, Paisani DM, Borges MC, Dantas BG, Caser EB, Victorino JA, Filho WO, Amato MBP, Cavalcanti AB. Driving Pressure-limited Strategy for Patients with Acute Respiratory Distress Syndrome. A Pilot Randomized Clinical Trial. Ann Am Thorac Soc. 2020 May;17(5):596-604. doi: 10.1513/AnnalsATS.201907-506OC. PMID 32069068